CLINICAL TRIAL: NCT07135206
Title: Perioperative Risk Assessment of Acute Kidney Injury Related to Pulmonary Endarterectomy Under Deep Hypothermic Circulatory Arrest
Brief Title: Risk of Acute Kidney Injury in Pulmonary Endarterectomy
Acronym: PEAAKI
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Li Fang Wang, Dr. Li Fang Wang, China-Japan Friendship Hospital
Other Study IDs: ZRYH-PEA-AKI-2025
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Venous blood (3mL per time point) and mid-stream urine (5mL per time point) will be collected. Serum and urine supernatant will be stored at -80℃ after centrifugation. Samples are used for detecting biomarkers such as NGAL and KIM-1, without DNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEA Patients with AKI Risk Assessment Cohort: This cohort integrates retrospective and prospective data from patients undergoing pulmonary endarterectomy (PEA) with deep hypothermic circulatory arrest (DHCA) at China-Japan Friendship Hospital. It includes: 1) Retrospective cases (2016-2025, ~240 cases) to explore perioperative risk factors for PEA-related acute kidney injury (AKI); 2) Prospective cases (2025-2027, 44 cases) to validate prediction models and analyze dynamic biomarkers (e.g., NGAL, KIM-1). The cohort aims to comprehensively assess AKI risk through combined analysis of historical and real-time data.

SUMMARY:
This study aims to assess the perioperative risk factors for acute kidney injury (AKI) in patients undergoing pulmonary endarterectomy (PEA) with deep hypothermic circulatory arrest (DHCA). By analyzing retrospective data (2016-2025) from approximately 240 PEA patients and prospectively enrolling 44 patients (2025-2027), we will identify clinical risk factors, establish and validate a comprehensive prediction model, and explore the dynamic characteristics and predictive value of novel biomarkers (e.g., NGAL, KIM-1). The goal is to improve early warning and management of PEA-related AKI, thereby enhancing patient outcomes.

DETAILED DESCRIPTION:
Background: PEA is the radical treatment for chronic thromboembolic pulmonary hypertension (CTEPH) and pulmonary artery sarcoma, requiring DHCA to ensure a bloodless surgical field. However, AKI occurs in 10-49% of PEA patients, significantly higher than neurological injury, leading to prolonged hospitalization and increased mortality. The risk factors and predictive biomarkers for PEA-related AKI remain unclear, highlighting the need for this research.

Study Design: A single-center, dual-cohort study including:

Retrospective Cohort: Patients who underwent PEA at China-Japan Friendship Hospital from 2016 to 2025. Data on baseline characteristics, intraoperative parameters (CPB/DHCA duration, perfusion pressure), postoperative renal function (based on KDIGO criteria), and outcomes (e.g., renal replacement therapy) will be collected to identify risk factors.

Prospective Cohort: Patients scheduled for PEA from 2025 to 2027. Clinical data and biological samples (blood/urine) will be collected at multiple time points (preoperatively, 2h/6h during CPB, 0h/24h/72h postoperatively) to measure biomarkers (NGAL, KIM-1, Scr, BUN). This cohort will validate the prediction model and assess biomarker performance.

Objectives:

Identify independent risk factors for PEA-related AKI. Develop and validate a perioperative prediction model for AKI. Clarify the dynamic changes and diagnostic/predictive value of novel biomarkers.

Outcome Measures:

Primary: AKI occurrence (KDIGO criteria). Secondary: AKI recovery rate, renal replacement therapy usage, hospital stay, 3-month mortality, and changes in renal/cardiopulmonary function.

Significance: This study will fill gaps in perioperative renal protection for PEA, provide an evidence-based risk assessment tool, and lay the foundation for optimized clinical management.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic thromboembolic pulmonary hypertension (CTEPH) or pulmonary artery sarcoma, and scheduled for or having undergone pulmonary endarterectomy (PEA) .

Aged 18 to 85 years . Underwent PEA using cardiopulmonary bypass (CPB) combined with deep hypothermic circulatory arrest (DHCA) technology .

Complete clinical data (including preoperative baseline data, intraoperative CPB/DHCA parameters, and postoperative respiratory, circulatory, and renal function data) .

Available renal function indicators at 3 months after surgery .

Exclusion Criteria:

Receiving preoperative maintenance renal replacement therapy . Complicated with severe liver failure, end-stage malignant tumors, or other diseases that affect short-term prognosis .

Missing key data (e.g., CPB/DHCA duration, postoperative 72-hour serum creatinine [Scr]) that cannot be supplemented .

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic thromboembolic pulmonary hypertension (CTEPH) or pulmonary artery sarcoma who undergo pulmonary endarterectomy (PEA) with deep hypothermic circulatory arrest (DHCA) at China-Japan Friendship Hospital. The study aims to evaluate perioperative risk factors for PEA-related acute kidney injury (AKI) and the value of novel biomarkers 。
Sampling Method: Non-Probability Sample
Enrollment: 284 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Acute Kidney Injury (AKI) after Pulmonary Endarterectomy (PEA) | Within 7 days after PEA surgery
  Acute kidney injury is defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria, which includes three stages based on serum creatinine (Scr) elevation and urine output reduction. Scr>1.5 times baseline or ≥0.3 mg/dl increase, or urine output <0.5 ml/kg/h for 6-12h

SECONDARY OUTCOMES:
Recovery of Renal Function | 1 months after surgery
  Proportion of patients whose Scr returns to ≤120% of baseline level before discharge.
Use of Renal Replacement Therapy (RRT) survey | Within 3 months after surgery
  Incidence of postoperative dialysis or continuous renal replacement therapy (CRRT).
duration of postoperative dialysis or continuous renal replacement therapy (CRRT). | Within 3 months after surgery
  Use of Renal Replacement Therapy (RRT)
Changes in Estimated Glomerular Filtration Rate (eGFR) from Baseline to 3 Months Postoperatively | 3 months after surgery
  This outcome assesses the numerical change in estimated glomerular filtration rate (eGFR) of patients from preoperative baseline to 3 months after surgery. eGFR will be calculated using a clinically validated formula (e.g., CKD-EPI formula), with the unit of mL/(min·1.73 m²).
Progression to Chronic Kidney Disease (CKD) at 3 Months Postoperatively | 3 months after surgery
  This outcome evaluates whether patients progress to chronic kidney disease (CKD) 3 months after surgery. CKD is defined as a persistent estimated glomerular filtration rate (eGFR) < 60 mL/(min·1.73 m²) for ≥ 3 months (meeting the standard CKD diagnostic criteria). The assessment result is a categorical variable (Yes/No) (i.e., whether the patient progresses to CKD).
Dynamic Changes of Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Kidney Injury Molecule-1 (KIM-1) and Their Correlation with AKI Occurrence and Severity | From preoperative to 72 hours postoperatively
  This outcome focuses on detecting the levels of two novel biomarkers-neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury molecule-1 (KIM-1)-in serum and urine samples collected from patients at multiple predefined time points. The sampling time points include the preoperative period, 2 hours and 6 hours during cardiopulmonary bypass (CPB), and 0 hours, 24 hours, and 72 hours postoperatively. Additionally, this outcome will analyze the correlation between the dynamic changes in NGAL and KIM-1 levels and two key indicators of AKI: the occurrence of AKI (as defined by KDIGO criteria) and the severity of AKI (KDIGO Stage I, II, or III). Biospecimens (3ml venous blood and 5ml midstream urine per time point) will be processed by centrifugation, with serum and urine supernatant stored at -80°C before biomarker detection, and no DNA extraction will be performed on the samples

CONTACTS AND LOCATIONS:
Overall Officials: Lifang Wang, M.D., Principal Investigator — China-Japan Friendship Hospital, Department of Anesthesiology
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with qualified researchers upon reasonable request, following publication of the study results. Shared data will include de-identified clinical information (baseline characteristics, intraoperative parameters, postoperative outcomes) and biomarker data, excluding direct identifiers to protect participant privacy. Data access will require approval from the institutional review board of China-Japan Friendship Hospital and a signed data use agreement specifying the purpose of use and confidentiality obligations. The data will be shared via a secure research data repository for up to 5 years after study completion
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data (IPD) and supporting information will be made available within 1 month after the publication of study results, with access maintained for 5 years after study completion.
Access Criteria: Eligible researchers must submit a research application specifying the purpose of data use and research plan, which will be reviewed and approved by the Institutional Review Board of China-Japan Friendship Hospital.A data use agreement must be signed, committing to use the data solely for scientific research, protect participants' privacy, refrain from unauthorized data transfer, and cite this study in published outcomes.De-identified data will be accessible through the hospital's designated secure data repository.
URL: https://www.medicalresearch.org.cn